CLINICAL TRIAL: NCT03553745
Title: How Body Awareness Promotes Mental Health During Yoga and Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Yoga Science Foundation (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Sara W Lazar, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017P001710
Record Dates: First submitted 2018-03-01; First posted 2018-06-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Negative Thoughts; Mild Depression; Stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gentle Yoga Program (Experimental): Program will meet twice a week for a 10-week period. Participants will be a part of gentle yoga sessions led by instructors specializing in the area.
  Interventions: Behavioral: Gentle Yoga Intervention
- Rigorous Yoga Program (Experimental): Program will meet twice a week for a 10-week period. Participants will be a part of rigorous yoga sessions led by instructors specializing in the area.
  Interventions: Behavioral: Rigorous Yoga Intervention
- Cardiovascular Exercise Program (Experimental): Program will meet twice a week for a 10-week period. Participants will be a part of cardiovascular exercise sessions led by instructors specializing in the area.
  Interventions: Behavioral: Physical Exercise Intervention

INTERVENTIONS:
Behavioral: Gentle Yoga Intervention — 10-week exercise program structured around gentle yoga practice.
  Arms: Gentle Yoga Program
Behavioral: Rigorous Yoga Intervention — 10-week exercise program structured around rigorous yoga practice.
  Arms: Rigorous Yoga Program
Behavioral: Physical Exercise Intervention — 10-week exercise program structured around cardiovascular exercise.
  Arms: Cardiovascular Exercise Program

SUMMARY:
The integrity of interoceptive networks is linked to resilience against depressive symptoms, whereas degradation of these networks is linked to apathy and deficits in emotion processing. The goal of this study is to compare two major styles of yoga and cardiovascular exercise through a 10-week training program to promote interoceptive awareness. The researchers hypothesize that improvement in affective symptomatology will be correlated with better interoceptive development. Changes in mood related symptoms and interoception will be assessed at baseline, week 12 and week 14, in a cohort of adults aged 18-55.

DETAILED DESCRIPTION:
A recent annual survey of U.S. college freshman has found consistently declining levels of emotional health over the past 25 years. Exposure to such stress can have profound longitudinal effects on well being, influencing risk for disease later in life. Physical exercise is linked to benefits across a variety of physical and psychological domains. While the affective and physiological consequences of exercise are well-documented, how they work to improve subjective well-being is unclear. It has been suggested that exercise promotes well-being by increasing interoception. The integrity of interoceptive networks is linked to resilience against depressive symptoms, whereas degradation of these networks is linked to apathy and deficits in emotion processing. The goal of this study is to compare two major styles of yoga and cardiovascular exercise through a 10-week training program to promote interoceptive awareness. The researchers hypothesize that improvement in affective symptomatology will be correlated with better interoceptive development. Changes in mood related symptoms and interoception will be assessed at baseline, week 12 and week 14, in a cohort of adults aged 18-55.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Have negative mood symptoms (depression, anxiety, stress)
* Is healthy and independent enough in daily life to attend study classes

Exclusion Criteria:

* Pregnant women or women who are planning to become pregnant during the study period
* History of structural brain disease, mass lesion, stroke, epilepsy
* History of addictive disorder or significant substance abuse
* Neurological disorders or reversible causes of dementia
* Suicidality or history of psychosis
* Currently attending regular yoga or aerobic exercise practice, or participated in more than 6 formal meditation, aerobic, or yoga classes in the past 12 months
* Self-reported cognitive impairment and other disorders which may preclude safe participation in the program including acute major depression, bipolar or severe personality disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Change in Interoceptive Acuity | 14 weeks
  Interoceptive acuity will be assessed at baseline, week 12 and week 14. Data collection at three time points will be used to assess changes in interoceptive acuity over the timeline.

SECONDARY OUTCOMES:
Peripheral Inflammatory Markers of Stress by collecting Dried Blood Spot (DBS) | 14 weeks
  Dried Blood Spot (DBS) will be collected at baseline, week 12 and week 14. This will be used to assess changes in levels of peripheral markers of inflammation (C-reactive protein, cytokines [IL-6]) in the blood as an indicator of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States